CLINICAL TRIAL: NCT01716546
Title: Phase I/II, Multicenter, Single-Arm Clinical Trial of Panitumumab in Combination With Cisplatin, Fluourouracil and Docetaxel (DCF) in Locally Advanced or Metastatic Cancer of the Stomach and Gastro-oesophageal Junction.
Brief Title: Trial of Panitumumab Cisplatin, Fluourouracil and Docetaxel in Locally Advanced or Metastatic Gastric Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Not reached the primary endpoint target according to the statistical design
Sponsor: Hellenic Oncology Research Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT/09.10
Record Dates: First submitted 2012-10-02; First posted 2012-10-30 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2015-10

CONDITIONS: Gastric Cancer
Keywords: Advanced cancer of the stomach; Chemotherapy - naive patients; DCF
MeSH Terms: conditions — Stomach Neoplasms | interventions — pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Panitumumab plus DCF
  Interventions: Drug: Pazopanib

INTERVENTIONS:
Drug: Pazopanib
  Other Names: Pazopanib: 800mg once a day for up to 2 years from date of first dose

SUMMARY:
Investigators propose to study the effect of panitumumab when combined with an active regimen, such as DCF (Docetaxel/Cisplatin/Fluourouracil), in previously untreated patients with advanced cancer of the stomach.

DETAILED DESCRIPTION:
Investigators propose a phase I/II study in order to evaluate the effect of panitumumab when combined with an active regimen, such as DCF (Docetaxel/Cisplatin/Fluourouracil), in chemotherapy - naive patients with advanced cancer of the stomach.

Investigators hypothesize that the addition of panitumumab to DCF regimen in advanced cancer of the stomach and gastroesophageal junction is feasible, well tolerated and could achieve an objective response rate of greater than 40%.

The 2-weekly schedule of DCF will be used as chemotherapy since a recently presented trial demonstrated a comparable efficacy but a more favourable toxicity profile comparable to the 3-weekly schedule.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven inoperable locally advanced or metastatic adenocarcinoma of the stomach (including adenocarcinoma of the gastrooesophageal junction)
* Patient's age between 20 and 70 years old
* Measurable disease defined by RECIST criteria
* Patients with non-measurable disease could be enrolled in the phase I part of the study
* ECOG performance status ≤ 1
* Hgb ≥ 8g/dL, WBC ≥ 3 x 109/L , neutrophils count ≥ 1.5 x 109/L , platelets ≥100 x 109/L, Creatinine clearance ≥50 mL/min, Total bilirubin ≤ 1.5 X UNL, AST, ALT and ALP ≤ 2.5 x UNL
* No prior chemotherapy or more than 6 months from adjuvant chemotherapy or chemo-radiation
* Estimated life expectancy more than 3 months
* Written informed consent

Exclusion Criteria:

* Gastrointestinal bleeding
* Clinically relevant, symptomatic excessive amounts of ascites resulting in patient's discomfort
* CNS metastases
* History of hypersensitivity to fluoropyrimidines, docetaxel or platinum compounds
* Any previous chemotherapy or radiotherapy for advanced disease
* Patient pregnant or breast feeding, or planning to become pregnant within 6 months after the end of treatment
* Patient (male or female) is not willing to use highly effective methods of contraception (per institutional standard) during treatment and for 6 months (male or female) after the end of treatment
* Known hypersensitivity reaction to the component of the treatment
* Active infection or malnutrition or bowel obstruction
* Legal incapacity or limited legal capacity
* Definite contraindications for the use of corticosteroids
* History of interstitial lung disease e.g. pneumonitis or pulmonary fibrosis or evidence of interstitial lung disease on baseline chest CT scan
* Chronic inflammation of the bowel
* Clinically significant cardiovascular disease (including myocardial infarction, unstable angina, symptomatic congestive heart failure, serious uncontrolled cardiac arrhythmia) ≤ 1 year before enrollment
* Medical or psychological condition which in the opinion of the investigator would not permit the subject to complete the study or sign meaningful informed consent
* A second primary tumor other than non-melanoma skin cancer or in situ cervical cancer

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2011-07; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Objective response rate | Every 8 weeks
  Patients will be followed for disease evaluation every eight (8) weeks from the first day of chemotherapy until the first documentation of disease progression

SECONDARY OUTCOMES:
Progression Free Survival | 1 year
  Patients will be evaluated from the date of the first chemotherapy cycle until the date of first documented progression or date of death from any cause, whichever came first
Overall Survival | 1 year
  Patients will be evaluated for overall survival from the date of the first chemotherapy cycle until the date of death from any cause
Maximum Tolerated Dose of the combination | Up to 4 weeks
  Patients will be evaluated for toxicity profil on Day 1 of the first two chemotherapy cycle (cycle repeated every 2 weeks)

CONTACTS AND LOCATIONS:
Locations (9):
- Greece (9):
  - "IASO" General Hospital of Athens, Athens
  - 401 Military Hospital of Athens, Athens
  - Air Forces Military Hospital of Athens, Athens
  - "Ag.Georgios" General Hospital of Chania, Chania
  - University Hospital of Crete, Dep of Medical Oncology Heraklion, Greece, Heraklion
  - State General Hospital of Larissa, Larissa
  - "Metaxa's" Anticancer Hospital of Piraeus, 1st Dep of Medical Oncology, Piraeus
  - "Theagenion" Anticancer Hospital of Thessaloniki, 2nd Dep of Medical Oncology, Thessaloniki
  - Diabalkaniko General Hospital of Thessaloniki, Thessaloniki